CLINICAL TRIAL: NCT01381510
Title: Establishing the Benefits of Adherence to Enlarged Prostate Treatment: A Validation Study Linking Adherence to Outcomes Using the Market Scan Database
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113909
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; Adherence; Acute urinary retention; Enlarged prostate; 5-alpha reductase inhibitor; Surgery; Cost and cost analysis
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — 5-alpha Reductase Inhibitors; Finasteride; Dutasteride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adherent BPH patients: Patients with benign prostatic hyperplasia (BPH) who are adherent to 5-alpha reductase inhibitor (5ARI) therapy based on a medication possession ratio (MPR). Analyses will be conducted with threshold adherence levels of 70%, 75% and 80%
  Interventions: Drug: 5-alpha Reductase Inhibitor (5ARI)
- Non-adherent BPH patients: Patients with BPH who are not adherent to 5ARI therapy based on an MPR and threshold levels of less than 70%, less than 75% and less than 80%
  Interventions: Drug: 5-alpha Reductase Inhibitor (5ARI)

INTERVENTIONS:
Drug: 5-alpha Reductase Inhibitor (5ARI) — A 5ARI: Either dutasteride or finisteride
  Other Names: Proscar ® (finasteride); Avodart ® (dutasteride)

SUMMARY:
Adherence and length of therapy with 5-alpha reductase inhibitor (5ARI) treatment may be associated with improved clinical outcomes of enlarged prostate (EP) as well as lower health care costs.

The objective of this retrospective database analysis is to quantify the relationship between adherence and length of therapy with a 5ARI and the likelihood of acute urinary retention (AUR) or prostate surgery (emergency and non-emergency) in patients with benign prostatic hyperplasia (BPH). The study will also measure the economic impact associated with these medical encounters.

The MarketScan database contains data from people with commercial health insurance and Medicare and includes both medical and pharmacy data that are sourced directly from health plans and employers. Approximately 18 million covered lives will be utilized for this study in the time period from January 1, 2003 to September 30, 2009.

This study is a retrospective cohort analysis of medical claims data.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 50 years or older
* A diagnostic claim of benign prostatic hyperplasia (International Classification of Diseases, Ninth Revision, Clinical Modification [ICD-9-CM] codes 222.2x or 600.xx)
* A prescription claim for a 5-alpha reductase inhibitor (5ARI) for at least 60 days during the observation period
* Continuous health plan eligibilitiy for 6 months prior to and at least 150 days after the initial 5ARI prescription

Exclusion Criteria:

* A diagnosis of prostate cancer (ICD-9-CM codes 185.xx, 198.82, 233.4, 236.5, 239.5, V10.46)
* A diagnosis of bladder cancer (ICD-9-CM codes 188.xx, 198.1, 223.3, 233.7, 239.4, V10.51),
* A procedure code for any prostate-related surgery prior to the index date or 150 days after the index date
* A diagnosis code for acute urinary retention (AUR) prior to the index date or 150 days after the index date

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is populated with claims data from male health plan members and Medicare patients age 50 and older who were continuously enrolled in a health plan that feeds into the MarketScan database between July 1, 2003 and May 1, 2009. Patient records were analyzed for 6 months prior to and at least 150 days following the index date for the first 5-alpha reductase inhibitor (5ARI) treatment
Sampling Method: Non-Probability Sample
Enrollment: 54459 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The occurence of a diagnosis code for acute urinary retention (AUR) or a procedure code for prostate surgery | One year following the first date of 5ARI therapy
  The occurence of a code for either AUR or prostate surgery will be identified for patients who were adherent with 5ARI therapy as measured with a medication possession ratio (MPR)

SECONDARY OUTCOMES:
Mean costs associated with AUR or prostate surgery | One year following the first date of 5ARI therapy
  The mean costs of outpatient and inpatient visits associated with the diagnosis code for AUR or the procedure codes for prostate surgery will be compared between patients who were compliant with 5ARI therapy and those who were not

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline